CLINICAL TRIAL: NCT02944903
Title: Lung Cancer Screening Practice in Chest Physicians
Brief Title: Audit of Lung Cancer Screening Practice in Chest Physicians: An Update
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aliae AR Mohamed Hussein, Prof. Dr. Aliae AR Mohamed-Hussein, Professor of Pulmonology, Assiut University
Other Study IDs: AssiutU2
Record Dates: First submitted 2016-10-23; First posted 2016-10-26 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Lung Cancer Screening
Keywords: audit; Lung cancer; screening practice; Egypt
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Audit — Questionnair

SUMMARY:
The investigators will conduct nationally representative survey in chest physicians in Egypt in 2016-2017. Self-administered questionnaire will be used to assess the physicians' knowledge of lung cancer screening guidelines, beliefs about the effectiveness of screening tests, and ordering of screening chest radiography, low-dose spiral computed tomography, or sputum cytology in the past 12 months.

DETAILED DESCRIPTION:
Although current practice guidelines do not recommend screening asymptomatic patients for lung cancer, physicians may still order lung cancer screening tests. No recent national survey of health care professionals has focused on lung cancer screening

ELIGIBILITY:
Inclusion Criteria:

* Physicians practising in Egypt (Chest physicians, general practitioners, and general internists)

Exclusion Criteria:

* Other nationalities
* Other specialities

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Chest physicians, general practitioners, and general internists
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2016-10; Primary Completion 2017-04 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Assessment of the use of guidelines of lung cancer screening | one year

SECONDARY OUTCOMES:
Self- administrated questionnaire | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Aliae Mohamed-Hussein, MD, Principal Investigator — Professor of Pulmonology- Faculty of Medicine-Assiut University
Locations (1):
- AssiutU, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided